CLINICAL TRIAL: NCT04985084
Title: Development and Testing of a Social Cognitive Theory-based Dietary Behavioral Intervention in Gastric Cancer Survivors: Protocol for a Pilot Randomized Controlled Trial
Brief Title: Development and Testing of a Social Cognitive Theory-based Dietary Behavioral Intervention in Gastric Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Dr CHENG Huilin, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 02
Record Dates: First submitted 2021-07-05; First posted 2021-08-02 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Stomach Neoplasms; Cancer Survivors
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): A 4-week dietary behavioral intervention provided by a registered nurse who has received nutrition training.
  Interventions: Behavioral: The intervention group
- Usual care (Other): General dietary advice provided by the ward nurses.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: The intervention group — The intervention will last for four weeks and target six dietary behaviors related to gastric cancer. The intervention components include one session of face-to-face education prior to discharge and three sessions of telephone counselling after discharge. The face-to-face education will last for 20 to 30 minutes and each session of telephone counselling will last for 10 to 20 minutes. All the interventional sessions are individual based.
  Arms: The intervention group
Other: Usual care — General dietary advice provided as routine by the ward nurses before discharge from the hospital.
  Arms: Usual care

SUMMARY:
This study aims to develop a Social Cognitive Theory (SCT)-based dietary behavioral intervention for gastric cancer survivors, and explore the feasibility, acceptability, and preliminary effectiveness of delivering this intervention. This study includes two phases: intervention development in phase 1 and a pilot randomized controlled trial (RCT) in phase 2.

During phase 1, the initial intervention protocol has been developed based on the SCT and literature review, which was further refined and/or enriched based on evidences from a qualitative descriptive study and an expert consultation. The qualitative descriptive study has been conducted from July to November 2021, and the expert consultation has been conducted from December 2021 to January 2022. For the qualitative descriptive study, purposive sampling was used to select eligible participants in patients who had a gastrectomy within two years from a tertiary hospital in Wuhan city, China. Three focus group interviews were performed with 13 participants via WeChat. Interviews were audio-recorded, transcribed verbatim, and analyzed using conventional qualitative content analysis. Data collection and analysis proceeded simultaneously until data saturation was reached. For the expert consultation, six experts majoring in nursing, digestive oncology, or nutrition were invited to assess the content validity of the intervention protocol. Data analysis of the qualitative descriptive study and the expert consultation is ongoing.

During phase 2, the pilot RCT for testing the feasibility, acceptability, and preliminary effectiveness of the proposed intervention is started. All participants are recruited through convenience sampling from a tertiary hospital in Wuhan city, China. Sample size of the pilot RCT is proposed to be 72. After randomization, the participants are assigned to one of two groups, either the intervention group, which receive a 4-week dietary behavioral intervention; or the control group, which receive usual care only. The 4-week dietary behavioral intervention targets six dietary behaviors related to gastric cancer and is delivered by a registered nurse who has received around 32 hours of nutrition training. The intervention includes one session of face-to-face education and three sessions of telephone counselling; all sessions are individual based. The usual care is general dietary advice provided by the ward nurses before discharge. The general dietary advice is provided orally and printed in the discharge plan. The primary outcomes are feasibility and acceptability. The secondary outcomes include dietary consumption, quality of life, and self-efficacy. Outcome measurements are conducted at baseline (before randomization), and week 5 (after intervention). Generalized estimating equation model analyses will be conducted to examine group-by-time interaction effects.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18 years or above；
* A confirmed diagnosis of gastric cancer (stage I-III)；
* Completed primary cancer treatments including surgery, and/or chemotherapy， and/or radiotherapy；
* Currently free of cancer；
* Able to read, write and speak Mandarin.

Exclusion Criteria:

* Unable to eat orally；
* With poor performance status as determined by the Eastern Cooperative Oncology Group (ECOG) scores ≥ 2;
* With poor cognitive status as determined by the Montreal Cognitive Assessment 5 minute Test <11;
* Taking part in other dietary interventions or under regular follow-up by a dietitian.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome: time to complete the recruitment | Immediately after completion of the intervention (T1)
  Time to complete the recruitment will be assessed by the time duration from the beginning to the completion of the recruitment.
Feasibility outcome: eligibility rate | Immediately after completion of the intervention (T1)
  Eligibility rate will be calculated by dividing the number of participants eligible by the number of participants screened.
Feasibility outcome: recruitment rate | Immediately after completion of the intervention (T1)
  Recruitment rate will be calculated by dividing the number of eligible participants who have consented and been randomized by the total number of eligible participants.
Feasibility outcome: retention rate | Immediately after completion of the intervention (T1)
  Retention rate will be calculated by dividing the number of participants completed the study with valid outcome data by the number of participants randomized.
Feasibility outcome: attendance rate | Immediately after completion of the intervention (T1)
  Attendance rate will be calculated by dividing the number of participants completed 4 interventional sessions by the number of participants assigned to the intervention group.
Acceptability outcome: participants' satisfaction and perspectives of the intervention | Immediately after completion of the intervention (T1)
  Participants' satisfaction and perspectives of the intervention will be assessed using a self-developed questionnaire designed for the study.

SECONDARY OUTCOMES:
Dietary consumption | Baseline before randomization (T0); Immediately after completion of the intervention (T1)
  Dietary consumption will be measured through telephone-assisted 24-hour dietary recall in three non-consecutive days (E.g., two workdays and one day during the weekend)
Health-related quality of life | Baseline before randomization (T0); Immediately after completion of the intervention (T1)
  Health-related quality of life will be assessed using the 46-item Functional Assessment of Cancer Therapy-Gastric (FACT-Ga) questionnaire. Each item is scored from 0 to 4 and the total score range from 0 to 184, with a higher score indicating better quality of life.
General self-efficacy | Baseline before randomization (T0); Immediately after completion of the intervention (T1)
  General self-efficacy will be assessed using the 10-item general self-efficacy scale. Each item is scored from 0 to 4 and the total score range from 0 to 40, with a higher score indicating higher general self-efficacy.
Dietary behavior self-efficacy | Baseline before randomization (T0); Immediately after completion of the intervention (T1)
  Dietary behavior self-efficacy will be assessed using a self-developed 6-item dietary behavior self-efficacy scale. Each item is scored from 0 to 4 and the total score range from 0 to 24, with a higher score indicating higher dietary behavior self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Huilin Cheng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gan T, Cheng H, Tse MYM, He N. Development of a nurse-led, evidence-based, and theory-informed dietary intervention to modify multiple unhealthy dietary behaviors in gastric cancer survivors. Asia Pac J Oncol Nurs. 2025 Jun 9;12:100739. doi: 10.1016/j.apjon.2025.100739. eCollection 2025 Dec. PMID 40611825